CLINICAL TRIAL: NCT05940285
Title: Evaluation of the Diagnostic Performance of Dynamic Myocardial Perfusion Scintigraphy in Comparison With Invasive Intracoronary FFR Measurement, in the Assessment of Significant Residual Coronary Stenosis After Acute Coronary Syndrome: Dyna-MI Pilot Study.
Acronym: Dyna-MI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC22_0698
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Myocardial Infarction
Keywords: Dynamic 99mTc-Tetrofosmin CZT-SPECT; Myocardial perfusion imaging; fractional flow reserve; acute coronary syndrome
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Experimental): Patients included in the study will undergo subsequently at 1-month after acute coronary syndrome Dynamic 99mTc-Tetrofosmin CZT-SPECT followed by FFR and IMR assessment
  Interventions: Diagnostic Test: Dynamic 99mTc-Tetrofosmin CZT-SPECT

INTERVENTIONS:
Diagnostic Test: Dynamic 99mTc-Tetrofosmin CZT-SPECT — Patients included in the study will undergo subsequently at 1-month after acute coronary syndrome Dynamic 99mTc-Tetrofosmin CZT-SPECT followed by FFR and IMR assessment

SUMMARY:
Dynamic 99mTc-Tetrofosmin CZT-SPECT myocardial perfusion imaging (MPI) is an advanced functional imaging technique giving important myocardial flow quantification added data in comparison with conventional MPI, especially in coronary multi vessel disease. A large-scale validation of diagnostic performances of myocardial flow reserve (MFR) estimated with Dynamic 99mTc-Tetrofosmin CZT-SPECT MPI would allow a non-invasive approach instead of invasive intra-coronary fractional flow reserve (FFR) measurement. The aim of this prospective study is to assess diagnostic performances of MFR calculated with dynamic 99mTc-Tetrofosmin CZT-SPECT MPI in comparison with invasive intra-coronary FFR measurement in patients with significant residual coronary arteries stenosis after acute coronary syndrome .

ELIGIBILITY:
Inclusion Criteria:

* Adult patient.
* Multi vessel coronary arteries disease (at least one non-culprit coronary stenosis >= 50%) diagnosis during

  * primary percutaneous coronary intervention < 12h after ST-elevation myocardial infarction opercutaneous revascularisation of the culprit lesion within 24 to 48 hours of an acute non-ST-segment elevation coronary syndrome.
* Written consent.
* Social security affiliation

Exclusion Criteria:

* Non adult patient.
* Adult patient under tutelage.
* Reproductive age women.
* Medical history of myocardial infarction or coronary artery bypass surgery.
* Cardiogenic shock.
* Cardiomyopathy.
* Regadenoson/adenosine/FFR contraindication.
* 99mTc-Tetrofosmin hypersensibility.
* Small non-culprit coronary arteries.
* Participation to another interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2027-10-20 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, predictive positive value, negative predictive value, accuracy of MFR in comparison with FFR | within one month after ST-elevation myocardial infarction
  To determine MFR diagnostic performances in comparison with FFR

SECONDARY OUTCOMES:
best MFR cut-off value | within one month after ST-elevation myocardial infarction
  To determine the best MFR cut-off value correlated with FFR value < 0.8
MFR value correlated with IMR | within one month after ST-elevation myocardial infarction
  analysis of discrepancies between MFR value correlated with IMR (if low MFR value and normal FFR value)
Sensitivity, specificity, predictive positive value, negative predictive value, accuracy of MFR in comparison with conventional static MPI | within one month after ST-elevation myocardial infarction
  To determine MFR diagnostic performances in comparison with conventional static MPI
Sensitivity, specificity, predictive positive value, negative predictive value, accuracy of QFR in comparison with FFR value | within one month after ST-elevation myocardial infarction
  QFR value at the index procedure in comparison with FFR value

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France